CLINICAL TRIAL: NCT01265849
Title: Phase III Study of LI [Multikine®] Plus SOC (Surgery + Radiotherapy or Surgery + Concurrent Radiochemotherapy) in Subjects With Advanced Primary Squamous Cell Carcinoma of the Oral Cavity/Soft Palate vs. SOC Only
Brief Title: Efficacy and Safety Study of Leukocyte Interleukin,Injection (LI) to Treat Cancer of the Oral Cavity
Acronym: IT-MATTERS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CEL-SCI Corporation (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry); Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS001P3; 2010-019952-35 (EudraCT Number)
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Results first posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Soft Palate
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Injections; Cyclophosphamide; Indomethacin; Zinc; Geritol; Surgical Procedures, Operative; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LI + CIZ + SOC (Experimental): LI plus CIZ (cyclophosphamide, indomethacin and zinc-multivitamins) was given as neoadjuvant therapy prior to standard of care (SOC).
  Interventions: Biological: LI; Drug: Cyclophosphamide; Drug: Indomethacin; Dietary Supplement: Zinc; Procedure: Surgery; Drug: Cisplatin; Radiation: Radiotherapy
- Standard of Care (SOC) only (Active Comparator): SOC for previously untreated SCCHN patients is currently surgery (with curative intent) followed by either radiotherapy or combined radiochemotherapy depending on the patient's risk status for recurrence as determined at surgery.
  Interventions: Procedure: Surgery; Drug: Cisplatin; Radiation: Radiotherapy
- LI + SOC (Experimental): LI was administered without CIZ to determine the contribution of CIZ to the effects of LI.
  Interventions: Biological: LI; Procedure: Surgery; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Biological: LI — LI 400 IU (2.0mL total daily) 1.0 mL peritumoral, 1.0 mL perilymphatic 5x weekly x3 consecutive weeks administered as neoadjuvant therapy prior to SOC, (surgery followed by radiation or concurrent radiochemotherapy with cisplatin 100 mg/m^2 intravenously x3) to determine if LI plus CIZ affects the 3-5 year overall survival.
  Other Names: Multikine; Leukocyte interleukin, injection
  Arms: LI + CIZ + SOC; LI + SOC
Drug: Cyclophosphamide — Cyclophosphamide was administered IV bolus (one time only) at a dose of 300mg/m^2 three days prior to beginning treatment with LI. Standard of care (SOC) for previously untreated squamous cell carcinoma of the head and neck is currently surgery followed by radiotherapy (60-70Gy in 30 to 35 fractions over 6 to 7 weeks) for higher risk subjects (subjects determined at surgery to have adverse features per the National Comprehensive Cancer Network (NCCN) guidelines, such as, positive surgical margins, 2 or more clinically positive nodes or extracapsular nodal spread, etc. that would pre-dispose them for higher risk of recurrence) radiotherapy is combined with concurrent chemotherapy (cisplatin 100mg/m^2 intravenously on day 1 of weeks 1, 4 and 7 of radiotherapy.
  Arms: LI + CIZ + SOC
Drug: Indomethacin — One 25mg capsule of indomethacin was self administered orally (BID) beginning on day one of LI treatment daily until the day before surgery.
  Arms: LI + CIZ + SOC
Dietary Supplement: Zinc — One capsule daily self administered beginning on day one of treatment with LI until one day before surgery
  Other Names: Multivitamins
  Arms: LI + CIZ + SOC
Procedure: Surgery — Excise tumor and nodes
Drug: Cisplatin — Cisplatin was administered 100mg/m^2 IV concurrent with radiotherapy. The chemotherapy agent (cisplatin 100mg/m^2) was administered intravenously on day 1 of weeks 1, 4 and 7 of radiotherapy.
Radiation: Radiotherapy — Total 60 to 70 Gy (2Gy per day) in 30 to 35 fractions over 6 to 7 weeks to subjects determined at surgery to be at lower risk for recurrence (per NCCN guidelines). For subjects determined at surgery to be at higher risk for recurrence due to having positive surgical margins, 2 or more clinically positive nodes or extracapsular nodal spread etc. (per NCCN guidelines), radiotherapy (as above) is combined with concurrent chemotherapy (cisplatin 100 mg/m^2) intravenously on day 1 of weeks 1, 4 and 7 of radiotherapy.

SUMMARY:
The purpose of this study was to determine whether LI administered in combination with cyclophosphamide, indomethacin and zinc in a multivitamin (CIZ) combination prior to standard of care therapy (surgery followed by radiotherapy or concurrent radiochemotherapy) is safe and will increase the overall survival of subjects with previously untreated locally advanced primary squamous cell carcinoma of the oral cavity or soft palate at a median of 3 to 5 years

DETAILED DESCRIPTION:
Head and neck carcinomas constitute about 5% of all cancers annually worldwide. In the US there are about 65,000 new cases annually. Ninety percent are squamous cell carcinoma of the head and neck (SCCHN). Approximately 2/3 of SCCHN patients present on their first visit with locally advanced disease. The median 3 year overall survival (OS) for these patients with existing standard of care (SOC) therapies - surgery followed by radiotherapy or concurrent radiochemotherapy - is estimated to be between 52 and 55%; the 5 year OS is approximately 43%. There are clearly many of SCCHN patients not well served by available modalities.

Regional intra or perilymphatic and/or intratumoral or peritumoral low dose cytokine therapy may have important therapeutic effects in SCCHN patients and constitute an additional anti-tumor mechanism of action different and distinct from current SOC. Leukocyte Interleukin Injection (LI) [Multikine] contains a defined mixture of naturally derived cytokines and chemokines with demonstrated safety and immunomodulatory activity in animals and in man in Phase I and Phase II clinical trials. LI is administered prior to SOC and in combination with low non-chemotherapeutic doses of cyclophosphamide, indomethacin, and zinc (CIZ) in studies with LI. The results of these studies indicate that the local/regional injection of mixed interleukins (LI) with CIZ prior to SOC can overcome local immunosuppression, break tumor tolerance to tumor antigens and allow for a sustainable and effective anti-tumor immune response.

LI was tested in this large, global, multinational Phase III clinical trial to develop definitive proof of its efficacy and safety in treating SCCHN. The trial is an open-label randomized multi-center controlled study of LI + CIZ + SOC in subjects with advanced primary SCCHN of the oral cavity/soft palate vs. SOC [the comparator arm]. OS is the primary efficacy endpoint.

ELIGIBILITY:
Inclusion Criteria (main):

* Untreated SCCHN of oral cavity (anterior tongue, floor of mouth, cheek)/soft palate, categories T1N1-2M0,T2N1-2M0,T3N0-2M0,T4N0-2M0 (T4 allowed only if invasion of mandible is negligible i. e. 5mm or less) scheduled for SOC
* Primary tumor and any positive node(s) measurable in 2 dimensions
* Normal immune function
* No immunosuppressives with 1 year of entry
* KPS>70/100
* Age>18
* Male or Female (non-pregnant)
* Life expectancy >6 months
* Able to take oral medication
* Able to provide informed consent

Exclusion Criteria (main):

* Subjects to be treated with other than SOC
* Tumor invasion of bone (also see inclusion criteria)
* Tumor classifications T1N0, T2N0, T4N3, any TN classification with M1
* Tumors in locations other than those specified in inclusion criteria
* Active peptic ulcer (or on full-dose therapeutic anti-coagulants)
* Prior resection of jugular nodes ipsilateral to tumor
* Acute or chronic viral, bacterial immune or other disease associated with abnormal immune function
* Subjects on hemodialysis or peritoneal dialysis; or having a history of
* History of asthma, allergy to fluoroquinolone antibiotics, congestive heart failure, or on hemodialysis or peritoneal dialysis
* Any condition that in the opinion of the investigator would cause the subject to be unable to participate or tolerate the protocol regimen
* Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Talor, PhD, Study Director — CEL-SCI Corporation
Locations (102):
- United States (5):
  - Simmons Cancer Institute at Southern Illinois University, Springfield, Illinois
  - Henry Ford Health System Henry Ford Hospital, Detroit, Michigan
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Medical College Of South Carolina MSC550, Charleston, South Carolina
  - VA Puget Sound Healthcare System & University of WA, Seattle, Washington
- HNO-Klinik der medizinischen Universitat Graz, Graz, Austria
- Belarus (2):
  - N.N. Alexandrov Research Istitute of Oncology and Medical Radiology, Lyasny, Minsk Oblast
  - Vitebsk Regional Oncology Dispensary, Vitebsk
- Bosnia and Herzegovina (4):
  - University Clinical Centre Tuzla, Trnovac, Tuzla
  - Clinical Center Banja Luka, Banja Luka
  - University Clinical Hospital Mostar, Mostar
  - Clinical Centre University of Sarejevo Clinic for ENT, Sarajevo
- Canada (3):
  - St. Josephs Healthcare Department of Surgery, Hamilton, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - CHU de Quebec - L'Hotel Dieu de Quebec, Québec
- Croatia (6):
  - CHC Osijek, Osijek
  - General Hospital Dr. Josip Bencevic, Slavonski Brod
  - CH Dubrava, Zagreb
  - Clinical Hospital Center Zagreb Kispaticeva 12, Zagreb
  - KBC Sestre Milosrdnice, Zagreb
  - KBC Zagreb, Zagreb
- ICL 6 avenue Bourgogne CS30519, Vandœuvre-lès-Nancy, France
- Hungary (6):
  - University of Debrecen Medical and Health Scioence Centre, Debrecen, Hajdú-Bihar
  - National institute of Oncology, Budapest, Rath Gyorgy
  - Semmelweis University, Budapest
  - University of Pecs Institute of Oncotherapy, Pécs
  - University of Szeged Dept of Oral and Maxillofacial Surgery, Szeged
  - Markusovsky Teaching Hospital, Szombathely
- India (11):
  - Bibi General Hospital and Cancer Centre, Malkapet, Andhra Pradesh
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Sujan Regional Cancer Hospital & Amravati Cancer Foundation, Amravati, Maharashtra
  - Government Medical College and Hospital, Aurangabad, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Curie Manavata Cancer Center, Mumbai, Naka Nashik
  - Searoc Cancer Center, Jaipur, Rajashlan
  - V.N. Cancer Center G. Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - Regional Cancer Center, Kerola, Thiruvananthapuram
  - Galaxy Cancer Center, Ghaziabad, Uttar Pradesh
- Israel (2):
  - Rambam Health Care Campus, Sha‘ar Ha‘Aliya, Saint Haifa
  - Rabin Medical Center, Petah Tikva, Tikva
- Italy (2):
  - National Tumor Institute of Italy, Naples
  - Ospedale S.G. Moscati Santissima Annunziata, Taranto
- Malaysia (2):
  - Dept of Head and Neck Surgery School of Medical Sciences Univ. Sains, Kuantan, Pulau Pinang
  - University Kabangsan Medical Center, Kuala Lumpur
- Poland (9):
  - Wojewodzki Szpital Specjalistyczny im Kopernika, Lodz, Ul Paderewskiego 4
  - Swietokrzyskie Centrum Onkologii, Kielce, Ul. Artwinskiego 3
  - Centrum Onkologi-Instytut im. Marie Sklodowskiej-Curie, Warsaw, Ul. Roentgena 5
  - Centrum Onkologii im. Prof. Lukaszcyka, Warsaw, Ul. Roentgena 5
  - ul. M. Sklodowskiej-Curie 24A, Bialystok
  - Szpital Specialistyczny im. Ludwika Rydgiera, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Klinika Otolarryngologii I Onkologii Laryngologicznej, Lublin
  - Weilkopolskie Centrum Onkologii Klinika Chirurgii Glowy Szye Onkologii Laryngologiczne, Poznan
  - Uniwersitecki Szpital Kliniczny Klinika Otolaryngologii Chirugii Glowy i Szxyi, Wroclaw
- Romania (2):
  - Regional Institute of Oncology IASI, Iași
  - Spital Clinic Judetean Mures, Târgu Mureş
- Russia (7):
  - Sverdlovsk Regional Cancer Center, Sverdlov, Ekaterinberg
  - Leningrad Regional Oncology Center, Saint Petersburg, Leningradskaya
  - Kursk Regional Clinical Oncology Dispensary, Kursk
  - Blokhin Cancer Research Center, Moscow
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Budget Institution of Healthcare of Omsk Region Clincal Oncology Dispensary, Omsk
  - Ryazan Clinical oncology Dispensary, Ryazan
- Serbia (8):
  - Serbia Clinic for ENT and Maxillofacial Surgery, Belgrade, Pasterova 14
  - Clincal Center Serbia Clinic for Oral and Maxillofacial Surgery, Belgrade
  - Faculty of Dental Medicine Clinic for Maxillofacial Surgery, Belgrade
  - Military Medical Academy Clinic for Maxillofacial Surgery, Belgrade
  - Clinical Center Nis center for Oncology, Niš
  - Clinic for Stomatology department for maxillofacial Surgery, Niš
  - Clinical center Vojvodina Clinic for ORL, Novi Sad
  - Clinical Centre Vojvodina Clinic for Maxillofacial Surgery, Novi Sad
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Madrid North Universitaro de Sanchinnaro, Madrid
  - Complejo Hospitalario Univ. de Santiago, Santiago de Compostela
  - Consorsio Hospital General Universitario de valencia, Valencia
- Sri Lanka (2):
  - National Cancer Institute Dept of Clinical Oncology & Radiotherapy, Colombo
  - Oncology Unit Teaching Hospital Karapitya, Galle
- Taiwan (9):
  - Kaohsiung Branch Chang Gung Memorial Hospital, Niaosong, Kaohsiung
  - National Cheng Kung University Hospital, Taipei, Tainan
  - National Taiwan Research Hospital, Chengshan, Taipei
  - Linkou Branch Chang Gung Memorial Hospital, Guishan, Taoyuan
  - Changua Christian Hospital, Chang-hua
  - Buddhist Tzu Chi General Hospital, Hualien Branch, Hualien City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Shin-Kong Wu Ho-Su Memorial Hospital, Taipei
- Khon Kaen University Dept of Otolaryngology, Nai Muang, Thailand
- Turkey (Türkiye) (2):
  - Haceteppe University Dept of Otolaryngology - Head and Neck Surgery, Ankara
  - Acibadem University Maslak Hospital ENT Department, Istanbul
- Ukraine (10):
  - Cherkasky Regional Oncological Dyspensary Dept. Head and Neck tumour, Cherkasy
  - Clinical Diagnostic Laboratory of Dnepropetrovsk Municipal Institution City Multidisciplinary Clinical Hospital No. 4, Dnipro
  - Donetsk Regional Antitumor Center, Donetsk
  - Grigoriev Institute for Medical Radiology of National Academy of Medical Science of Ukraine Dept. of Remote, Combined Radiation and Complex Therapy, Kharkiv
  - Kharkiv Regional Clinical Oncology Center Dept. Of Head and Neck Tumour, Kharkiv
  - Kiev City Clinical Oncology Center of the Main Health Care Dept of Kiev Day Hospital Radiotherapy Dept., Kiev
  - Kiev City Clinical Oncology Center of the Main Health Care Dept. of the Kiev Day Hospital, Kiev
  - Lviv State OncologyRegional treatment and Diagnostic Center, Lviv
  - Sumy Regional Clinical Oncology Dyspensary, Sumy
  - Zaporiz'ka Regional Clinical Oncology Dispensary, Zaporiz'ka Oblast'
- Aintree University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan

REFERENCES:
- [Derived] Talor E, Timar J, Lavin P, Cipriano J, Markovic D, Ladanyi A, Karpenko A, Bondarenko I, Stosic S, Sobat H, Zhukavets A, Imamovic N, Chien CY, Bankowska-Wozniak M, Kisely M, Jovic R, Young JEM, Hao SP. Neoadjuvant leukocyte interleukin injection immunotherapy improves overall survival in low-risk locally advanced head and neck squamous cell carcinoma -the IT-MATTERS study. Pathol Oncol Res. 2025 Mar 21;31:1612084. doi: 10.3389/pore.2025.1612084. eCollection 2025. PMID 40191245
- See also: Click here for more information about this study: Phase 3 Efficacy and Safety Study of Leukocyte Interleukin,Injection (LI) to Treat Cancer of the Oral Cavity (IT-MATTERS) — http://www.cel-sci.com

RESULTS

PARTICIPANT FLOW:
Groups:
- LI + CIZ + SOC: LI plus CIZ (cyclophosphamide, indomethacin and zinc) is given as adjuvant therapy prior to standard of care (SOC).
- Standard of Care (SOC): SOC for previously untreated SCCHN patients is currently surgery followed by either radiotherapy or combined radiochemotherapy depending the patient's risk status for recurrence determined at surgery.
- LI + SOC: LI is administered without CIZ to determine the contribution of CIZ to the effects of LI.
Period: Overall Study
Arm/Group | LI + CIZ + SOC | Standard of Care (SOC) | LI + SOC
Started | 396 | 398 | 134
Completed | 350 | 337 | 115
Not Completed | 46 | 61 | 19
Not completed — Randomized//Treatment not initiated | 1 | 4 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Lost to Follow-up | 18 | 15 | 5
Not completed — Not otherwise specified | 1 | 6 | 1
Not completed — Withdrawal by Subject | 25 | 34 | 13

BASELINE CHARACTERISTICS:
Population: Five randomized subjects were excluded due to the Crimean war (4 cases could not be followed) and one USA case where the Principal Investigator did not sign the full CRF, which left 923 ITT subjects in the study.
Groups:
- LI + CIZ + SOC: LI plus CIZ (cyclophosphamide, indomethacin and zinc) is given as neoadjuvant therapy prior to standard of care (SOC).
- Standard of Care (SOC): SOC for previously untreated SCCHN patients is currently surgery followed by either radiotherapy or combined radiochemotherapy depending the patient's risk status for relapse determined at surgery.
- Total: Total of all reporting groups
Arm/Group | LI + CIZ + SOC | Standard of Care (SOC) | LI + SOC | Total
Number analyzed (Participants) | 395 | 394 | 134 | 923
Age, Continuous [Mean (Full Range); unit: years] | 56.5 [26 to 82] | 56.9 [22 to 84] | 55.9 [20 to 86] | 56.6 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 79 | 29 | 191
  Male | 312 | 315 | 105 | 732
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 190 | 186 | 57 | 433
  Unknown or Not Reported | 205 | 208 | 77 | 490
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 79 | 76 | 25 | 180
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 311 | 317 | 108 | 736
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Malaysia | 2 | 2 | 1 | 5
  Philippines | 1 | 1 | 0 | 2
  Taiwan | 17 | 16 | 7 | 40
  Thailand | 1 | 1 | 0 | 2
  India | 37 | 38 | 11 | 86
  Israel | 2 | 3 | 1 | 6
  Sri Lanka | 20 | 19 | 7 | 46
  Bosnia and Herzegovina | 16 | 18 | 6 | 40
  Serbia | 78 | 79 | 26 | 183
  Turkey | 1 | 0 | 0 | 1
  Belarus | 20 | 19 | 7 | 46
  Russia | 76 | 76 | 26 | 178
  Ukraine | 68 | 67 | 23 | 158
  Canada | 1 | 1 | 1 | 3
  Croatia | 23 | 24 | 8 | 55
  France | 1 | 0 | 0 | 1
  Hungary | 9 | 9 | 3 | 21
  Poland | 20 | 20 | 6 | 46
  Romania | 1 | 1 | 0 | 2
  United States | 1 | 0 | 1 | 2
Primary Tumor Location [Count of Participants; unit: Participants]
  Cheek (Buccal Mucosa) | 53 | 55 | 18 | 126
  Floor of Mouth | 111 | 116 | 37 | 264
  Oral Tongue | 182 | 178 | 63 | 423
  Soft Palate | 49 | 45 | 16 | 110
Tumor Code [Count of Participants; unit: Participants]
  T1: Tumor < 2 cm in greatest dimension | 21 | 12 | 4 | 37
  T2: Tumor > 2 and < 4 cm in greatest dimension or extension to lingual surface of epiglottis | 94 | 95 | 28 | 217
  T3: Tumor more than 4 cm in greatest dimension | 163 | 191 | 68 | 422
  T4a: Moderately advanced local disease | 117 | 96 | 34 | 247
Number of Nodes Involved [Count of Participants; unit: Participants]
  Missing | 1 | 0 | 0 | 1
  N0 | 190 | 180 | 62 | 432
  N1 | 108 | 118 | 37 | 263
  N2 | 96 | 96 | 35 | 227
TNM Stage [Count of Participants; unit: Participants] — Staging by the American Joint Committee on Cancer (AJCC). Baseline Tumor-Node-Metastasis (TNM) Stage: Tumors that are T1-T4 by the TNM classification system are included in the study. Nodal involvement (count) must be N0-N2 and no metastatic disease (M0).
  TNM Stage III includes T1N1M0, T2N1M0, T3N0M0, and T3N1M0.
  TNM Stage IV includes all with N2 or T4 (T1N2M0, T2N2M0, T3N2M0, T4N0M0, T4N1M0, T4N2M0.
  Stage IV A is is associated with a poorer (worse) prognosis than Stage III.
  Participants
    TNM Stage III | 218 | 228 | 75 | 521
    TNM Stage IV | 177 | 166 | 59 | 402

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was assessed using Kaplan-Meier life-table using a log rank test and confirmed further with tumor stage, tumor location, and geographic stratified log rank test. Both Stratified and unstratified log rank test are presented with the unstratified log rank test constituting the primary analysis. A two-sided p-value of 0.05 or less was considered statistically significant for comparing the two groups (i.e., Study comparator arms: LI+CIZ+SOC vs. SOC alone). Interim analyses were performed (by the iDMC) periodically throughout the study to assess safety, sample size and futility.
Time Frame: From the date of treatment assignment to death or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 395 | 134 | 394
months | 46.3 [39.3 to 55.0] | 58.1 [41.4 to 68.2] | 52.9 [46.5 to 66.6]
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); The primary objective was to compare overall survival in the LI + CIZ + SOC group to that in the SOC alone group for superiority of the former; Test type: Superiority; p = 0.4051, Log Rank — For the primary efficacy measure a two-sided p-value of 0.05 or less is considered to be statistically significant in comparing the LI+CIZ+SOC treatment vs. SOC alone for superiority; Log Rank statistic is based on an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.5402, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4128, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.89 to 1.32] — A Hazard Ratio < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.7181, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.9480, Log Rank; This log Rank p-value is based on a stratified analysis
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6101, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.81 to 1.42] — A hazard Ratio < 1.0 would favor LI + SOC

2. Primary Outcome: OS in Low Risk Subjects
Description: OS was assessed using Kaplan-Meier life-table using a log rank test and confirmed further with tumor stage, tumor location, and geographic stratified log rank test. Both Stratified and unstratified log rank test are presented with the unstratified log rank test constituting the primary analysis. A two-sided p-value of 0.05 or less was considered statistically significant for comparing the two groups (i.e., Study comparator arms: LI+CIZ+SOC vs. SOC alone). Low-risk assessment and data analysis was never performed during the study and was done only after database lock.
Time Frame: as for outcome 1
Population: Low Risk Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
months | 101.7 [64.1 to 101.7] | 68.2 [44.7 to NA] — The upper limit for the 95% Confidence Interval cannot be estimated, "Too few events ". | 55.2 [48.0 to NA] — The upper limit for the 95% Confidence Interval cannot be estimated, "Too few events".
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0478, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0137, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0236, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.48 to 0.95] — A Hazard Ratio < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4115, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.2862, Log Rank; This Log Rank statistic is based on a stratified analysis; This HR is presented as (LI + SOC) / SOC. A HR < 1.0 favors LI+SOC. Wald p-value for this HR is 0.3859
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.3859, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.52 to 1.29] — A Hazard Ratio < 1.0 would favor LI + SOC

3. Secondary Outcome: Local Regional Control (LRC)
Description: LRC is defined as the number of months from randomization to the date of documented local or regional failure (recurrence or progression) or date of last follow-up or death. LRC failure includes the reappearance (recurrence) of disease (at the original tumor sites), progressive disease (but not distant metastases), or any new disease (including new disease in lymph nodes), above the clavicle, not present at baseline. This is the traditional RTOG measure of local-regional control, also referred to as Freedom from Local Progression.
Time Frame: From the date of treatment assignment to LRC or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 395 | 134 | 394
months | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event. | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event. | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event.
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); The secondary endpoint LRC failure is analyzed similar to the primary OS endpoint. The primary comparison is LI+CIZ+SOC vs SOC; LI+SOC vs SOC results are also reported; Test type: Superiority; p = 0.7304, Log Rank — P-values are not adjusted for multiple comparisons; This Log Rank P-value is based on an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.7171, Log Rank — P-values are reported unadjusted for multiplicity; The Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.8020, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.79 to 1.36] — A Hazard Ratio < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4231, Log Rank; The Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6998, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.3944, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.81 to 1.69] — A Hazard Ratio < 1.0 would favor LI + SOC

4. Secondary Outcome: LRC in Low Risk Subjects
Description: LRC is defined as the number of months from randomization to the date of documented local or regional failure (recurrence or progression) or date of last follow-up or death. LRC failure includes the reappearance (recurrence) of disease (at the original tumor sites), progressive disease (but not distant metastases), or any new disease (including new disease in lymph nodes), above the clavicle, not present at baseline. This is the traditional RTOG measure of local-regional control, also referred to as Freedom from Local Progression. Low risk assessment and data analysis was never performed during the study and was done only after database lock.
Time Frame: From the date of treatment assignment to LRC or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Low Risk Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
months | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event. | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event. | NA [NA to NA] — Too few events occurred to estimate the median (95% CI) time-to-event.
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6142, Log Rank; The Log Rank statistic is based on an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.3024, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.42082, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.55 to 1.28] — A Hazard Ratio < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.9784, Log Rank; The Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.8461, Log Rank — This Log Rank statistic is based on a stratified analysis
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.8131, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.53 to 1.65] — A Hazard Ratio of < 1.0 would favor LI + SOC

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the number of months from randomization to the date of first documented, progressive disease (any tumor recurrence, any new disease above clavicle or distant metastases) or the date of last follow-up or death. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest dimension (LD) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From the date of treatment assignment to PFS or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Intent to Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 395 | 134 | 394
months | 32.4 [25.5 to 43.4] | 37.0 [19.4 to 57.4] | 45.5 [23.5 to 51.2]
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); This secondary endpoint PFS is analyzed similar to OS and LRC; Test type: Superiority; p = 0.3303, Log Rank; This Log Rank statistic is from an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6669, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.3728, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.31] — A Hazard Ratio < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.5739, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.8162, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4728, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.84 to 1.43] — A Hazard Ratio < 1.0 would favor LI + SOC

6. Secondary Outcome: PFS in Low Risk Subjects
Description: PFS is defined as the number of months from randomization to the date of first documented, progressive disease (any tumor recurrence, any new disease above clavicle or distant metastases) or the date of last follow-up or death. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest dimension (LD) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions. Low risk assessment and data analysis was not performed during the study and was performed only after database lock.
Time Frame: From the date of treatment assignment to PFS or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Low Risk Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- LI + SOC: LI is administered without CIZ to determine the contribution of CIZ to the effects of CIZ.
- Standard of Care (SOC): SOC for previously untreated SCCHN patients is currently surgery followed by either radiotherapy or combined radiochemotherapy.
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
months | 66.4 [47.5 to 101.7] | 68.2 [37.0 to 112.4] | 51.5 [42.5 to 72.2]
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.1797, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 2: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0159, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0896, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.55 to 1.04] — A Hazard Ratio of < 1.0 would favor LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.5175, Log Rank; This Log Rank statistic is based on an unstratified analysis
Statistical Analysis 5: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4530, Log Rank; This Log Rank statistic is based on a stratified analysis
Statistical Analysis 6: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4376, Regression, Cox; The Cox Proportional Hazards Model included terms for treatment, tumor stage, tumor location, and geographic region; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.54 to 1.30] — A Hazard Ratio < 1.0 would favor LI + SOC

7. Secondary Outcome: Quality of Life by EORTC QLQ-C30 Global Health Status [GHS] at Month 2
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionaire C-30 Version 3.0 (EORTC QLQ-C30) V3.0 is composed of both multi-item scales and single-item measures. The Global Health Scale/QoL multi-item scale [GHS] is a comprised of two Items: Item 29 "How would you rate your overall health during the past week?", and item 30: "How would you rate your overall quality of life during the past week?". Both items are 7 point scales ranging from a score of 1 (very poor) to 7 (Excellent). The GHS is constructed by averaging Items 29 and 30 to obtain a raw score (RS). The RS is then transformed to a 0-100 scale by the equation GHS=100*[(RS-1)/6]. A higher score represents a higher ("better") QoL. Change in GHS is calculated as Observed - Baseline, so a positive change in GHS is improved QoL. Treatment comparisons are active treatment arms minus SOC, so a positive difference favors active treatment.
Time Frame: Global Health Status (GHS) at Baseline [pre-randomization], Long Term Follow-up Month 2
Population: Overall number of participants analyzed is the total number of subjects in the longitudinal model.
  The number of participants analyzed is the number of subjects assessed at each visit.
  This study is not powered for quality of life comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (0-100)
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 117 | 37 | 119
units on a scale (0-100) | 0.28 (1.82) | 7.95 (3.03) | 3.29 (1.83)
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Approximately 30% of participants completed the QOL instrument at first administration (Month2), thus the study did not have the power for QoL comparisons. These completer analyses are descriptive only; Test type: Superiority; p = 0.2100, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up at Month 2 is not adjusted for multiplicity; RMANCOVA with fixed stratification factors, trt, visit, trt*visit, and baseline, with a compound symmetry correlation structure; Mean Difference (Net) = -3.00, Standard Error of Mean 2.395 — Positive value for the difference (Mean Difference (Net)) favors LI + CIZ + SOC
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Approximately 30% of participants completed the QOL instrument at last administration (Month 36), thus the study did not have power for QoL comparisons. These completer analyses are descriptive only; Test type: Superiority; p = 0.1701, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up at Month 2 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = 4.67, Standard Error of Mean 3.401 — Positive value for the difference (Mean Difference (Net)) favors LI + SOC

8. Secondary Outcome: Quality of Life by EORTC QLQ-C30 Global Health Status [GHS] at Month 36
Description: as for outcome 7
Time Frame: Global Health Status (GHS) at Baseline [pre-randomization], Long Term Follow-up Month 36
Population: Overall number of participants analyzed is the total number of subjects with data at this visit.
  The number of participants analyzed is the number of subjects assessed at each visit.
  This study is not powered for quality of life comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (0-100)
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 112 | 44 | 119
units on a scale (0-100) | 7.64 (1.82) | 10.79 (2.85) | 6.33 (1.80)
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); LI + CIZ + SOC, Standard of Care (SOC); Test type: Superiority — This p-value for Long Term Follow-up at Month 36 is not adjusted for multiplicity; p = 0.5871, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Median Difference (Net) = 1.3, Standard Error of Mean 2.397 — Positive value for the difference (Mean Difference (Net)) favors LI + CIZ + SOC
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.1700, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = 4.46, Standard Error of Mean 3.247 — Positive value for the difference (Mean Difference (Net)) favors LI + SOC

9. Secondary Outcome: EORTC Quality of Life Questionnaire (QLQ) - Head & Neck Cancer Module: QLQ-H&N35 at Month 2
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionaire C-30 Version 3.0 supplementary Head & neck cancer module (EORTC QLQ-C30 - QLQ H&N35) items 1-4 make up the symptom score for pain, items 5-8 for swallowing. The 4 pain questions score: "pain in your mouth, pain in your jaw, soreness in your mouth, a painful throat?" The 4 swallowing questions score "problems swallowing: liquids, pureed food, solid food, choking? Item are scored as 1 (Not at all) to 4 (Very much). Each symptom scale is constructed by averaging the 4 items to obtain a raw score (RS). The RS is then transformed to a 0-100 scale by the equation symptom score (pain or swallowing)=100*[(RS-1)/3]. A high score for these symptom scales represents a high level of symptoms.Change in symptom is calculated as Observed - Baseline, so a negative change is reduced symptomatology . Treatment comparisons are active treatment arms minus SOC, so a negative difference favors active treatment.
Time Frame: Baseline [pre-randomization], Long Term Follow-up Month 2
Population: Overall number of participants analyzed is the total number of subjects in data at that visit.
  The number of participants analyzed is the number of subjects assessed at each visit.
  This study is not powered for quality of life comparisons.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (0-100)
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 117 | 37 | 120
units on a scale (0-100)
  Change from Baseline in Head & Neck PAIN at Long Term Follow-up Month 2 | -2.75 (1.66) | -2.80 (2.77) | -3.81 (1.67)
  Change from Baseline in Head & Neck SWALLOWING at Long Term Follow-up Month 2 | 8.11 (1.88) | 6.29 (3.13) | 7.31 (1.89)
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6296, Repeated Measures ANCOVA (RMANCOVA) — This p-value for head and neck pain at Long Term Follow-up Month 2 is not adjusted for multiplicity; RMANCOVA with fixed effects of treatment, visit, treatment by visit, tumor location & stage, geographic region, and baseline with compound symmetry; Mean Difference (Net) = 1.05, Standard Error of Mean 2.183 — Negative value for the difference (Mean Difference (Net)) favors LI + CIZ + SOC
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.7454, Repeated Measures ANCOVA (RMANCOVA) — This p-value for head and neck pain at Long Term Follow-up Month 2 is not adjusted for multiplicity; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 1.01, Standard Error of Mean 3.103 — Negative value for the difference (Mean Difference (Net)) favors LI + SOC
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.7452, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for swallowing at month 2 is not adjusted for multiplicity; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 0.80, Standard Error of Mean 2.465 — Negative value for the difference (Mean Difference (Net)) favors LI + CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.7710, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for swallowing at Month 2 is not adjusted for multiplicity; RMANCOVA with fixed effects of treatment, visit, treatment by visit, and baseline with compound symmetry; Mean Difference (Net) = -1.02, Standard Error of Mean 3.496 — Negative value for the difference (Mean Difference (Net)) favors LI + SOC

10. Secondary Outcome: EORTC Quality of Life Questionnaire (QLQ) - Head & Neck Cancer Module: QLQ-H&N35 at Month 36
Description: as for outcome 9
Time Frame: Baseline [pre-randomization], Long Term Follow-up Month 36
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale (0-100)
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 112 | 44 | 120
units on a scale (0-100)
  Change from Baseline in Head & Neck PAIN at Long Term Follow-up Month 36 | -9.47 (1.66) | -8.63 (2.61) | -8.42 (1.64)
  Change from Baseline in Head & Neck SWALLOWING at Long Term Follow-up Month 36 | 6.90 (1.89) | 1.66 (2.96) | 8.94 (1.86)
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.6337, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for head and neck pain at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -1.04, Standard Error of Mean 2.185 — Negative value for the difference (Mean Difference (Net)) favors LI + CIZ + SOC
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.9450, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for head and neck pain at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -0.20, Standard Error of Mean 2.962 — Negative value for the difference (Mean Difference (Net)) favors LI + SOC
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.4071, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for Swallowing at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -2.04, Standard Error of Mean 2.465 — Negative value for the difference (Mean Difference (Net)) favors LI+ CIZ + SOC
Statistical Analysis 4: Comparison: LI + SOC vs Standard of Care (SOC); Test type: Superiority; p = 0.0296, Repeated Measures ANCOVA (RMANCOVA) — This p-value for Long Term Follow-up for Swallowing at Month 36 is not adjusted for multiplicity; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -7.29, Standard Error of Mean 3.347 — Negative value for the difference (Mean Difference (Net)) favors LI + SOC

11. Secondary Outcome: Statistical Comparisons of Time-to-event Outcomes (OS, LRC, PFS) Were Repeated for Varying Levels of Histopathology (HP) Markers in Low Risk Subjects
Description: HP analysis was performed in a blinded manner by a central pathology laboratory at the end of the study on available samples. To examine potential effects of HP markers on time-to-event efficacy outcomes (OS, LRC, PFS), participants were classified by HP marker levels: 20 HP markers were classified as (low, medium, high), 2 HP ratios as (low, medium, high) and 14 HP combinations as (low, high), resulting in 94 (20*3+2*3+2*14) possible treatment comparisons of LI + CIZ + SOC to SOC. A total of 282 (94 x 3 efficacy outcomes) statistical tests (Cox proportional hazards regressions to test for a significant treatment effect in the model) were made. Significance (two-sided p<0.05 favoring LI + CIZ + SOC) were reported under LI + CIZ + SOC. Significant test results favoring SOC were reported under SOC. The total number of statistical comparisons between LI + CIZ + SOC and SOC (282) is reported under both arms.
Time Frame: From the date of treatment assignment to event (LRC,PFS,OS) or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: The analysis population is the Low Risk Intent to treat Population who had HP marker levels assessed and were in either treatment arm LI + CIZ + SOC or SOC. This includes 82 subjects in LI + CIZ + SOC and 95 subjects in standard of care (SOC). No statistical comparisons were made for the 33 Low Risk subjects with HP markers in treatment arm LI + SOC. No data were collected for this Outcome Measure for treatment arm LI + SOC..
Measure: Number; unit: N of Statistically Significant Results
Units Other Than Participants: Number of statistical tests
Arm/Group | LI + CIZ + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 82 | 95
Number analyzed (Number of statistical tests) | 282 | 282
N of Statistically Significant Results | 61 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Treatment comparisons of LI+CIZ+SOC v. SOC were repeated at all levels of HP, HP ratios, and HP combinations for endpoints OS, PFS, and LRC. Significant outcomes for the treatment term in the model (two-sided p<0.05) were accumulated; Test type: Superiority — Statistical tests were for a significant treatment effect in the Cox Proportional Hazards model including treatment, disease stage, tumor location, and geographical region; p < 0.05, Regression, Cox — Under the null hypothesis of no effect the expected number of significant test results would be balanced between treatments. The expected number (%) of statistically significant results would be approximately 14 (5%) of 282; % of significant test results = 21.6, 95% CI 2-sided [17.0 to 26.9]

12. Post Hoc Outcome: Tumor Response by RECIST 1.0
Description: Tumor response is evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) and confirmed by pathology at surgery. For target lesions as assessed by MRI or CT: Complete Response (CR) is disappearance of all target and non-target lesions, no new tumors, and normalization of tumor marker level. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions taken as a reference the baseline sum of LDs, and no new tumors. Objective response = CR + PR. Response was assessed to LI treatment and compared to controls (SOC) from randomization to surgery in the ITT population for recurrence.
Time Frame: From treatment assignment to planned surgery, 29-38 days for LI treated groups and as soon as practicable with within 8 - 38 days for the SOC group (median 33 days).
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 395 | 134 | 394
participants
  Complete Response (CR) | 5 | 0 | 0
  Partial Response (PR) | 27 | 13 | 0
  Objective Response (CR+PR) | 32 | 13 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); Null hypothesis is that percent (%) of participants with an objective response (CR+PR) is the same for LI + CIZ + SOC and SOC; Test type: Superiority; p < .0001, Fisher Exact; Percent (%) of Participants = 8.1, 95% CI 2-sided [5.6 to 11.2]
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Null hypothesis is that percent (%) of participants with an objective response (CR+PR) is the same for LI + SOC and SOC; Test type: Superiority; p < 0.0001, Fisher Exact; Percent (%) of Participants = 9.7, 95% CI 2-sided [4.7 to 14.7]

13. Post Hoc Outcome: Tumor Response by RECIST 1.0 in Low Risk Subjects
Description: Tumor response was evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). For target lesions as assessed by MRI or CT: Complete Response (CR) is disappearance of all target and non-target lesions, no new tumors, and normalization of tumor marker level. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions taken as a reference the baseline sum of LDs, and no new tumors. Objective response = CR + PR. Response was assessed to LI treatment and compared to controls (SOC) from randomization to surgery in the lower risk ITT population for recurrence.
Time Frame: as for outcome 12
Population: Low Risk Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
Participants
  Complete Response (CR) | 5 | 0 | 0
  Partial Response (PR) | 19 | 10 | 0
  Objective Response (CR+PR) | 24 | 10 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs Standard of Care (SOC); [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, Fisher Exact; Percent (%) of Participants = 15.2, 95% CI 2-sided [9.6 to 20.8]
Statistical Analysis 2: Comparison: LI + SOC vs Standard of Care (SOC); Null hypothesis is that percent (%) of participants with an objective response (CR+PR) is the same for LI + SOC and SOC; Test type: Superiority; p < 0.0001, Fisher Exact; Percent (%) of Participants = 18.5, 95% CI 2-sided [8.2 to 28.9]

14. Post Hoc Outcome: Survival by Objective Response (CR+PR)
Description: Survival is assessed as dead or alive at last follow-up. Tumor response is evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). For target lesions as assessed by MRI or CT: Complete Response (CR) is disappearance of all target and non-target lesions, no new tumors, and normalization of tumor marker level. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions taken as a reference the baseline sum of LDs, and no new tumors. Objective response = CR + PR.
Time Frame: Objective Response: from treatment assignment to surgery: 29-38 days for LI-treated & 8-38 days for SOC (median 33 days). Survival from treatment assignment to death or the last follow-up date. Maximum follow-up was approximately 113 months.
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 395 | 134 | 394
Participants
  Non-responder and Alive | 166 | 56 | 204
  Non-responder and Dead | 197 | 65 | 190
  Responder and Alive | 25 | 10 | 0
  Responder and Dead | 7 | 3 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC; The null hypothesis that survival is unrelated to objective response versus the alternative hypothesis that objective response is predictive of increased survival for participants receiving LI + CIZ + SOC; Test type: Superiority; p = 0.0007, Fisher Exact
Statistical Analysis 2: Comparison: LI + SOC; The null hypothesis is that survival is unrelated to objective response versus the alternative that response is predictive of increased survival in subjects receiving LI + SOC; Test type: Superiority; p = 0.0434, Fisher Exact
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs LI + SOC; The null hypothesis is that survival is unrelated to objective response versus the alternative hypothesis that objective response is predictive of increased survival for participants receiving LI, considering both treatment groups combined; Test type: Superiority; p < 0.0001, Fisher Exact

15. Post Hoc Outcome: Survival by Objective Response (CR+PR) in Low Risk Subjects
Description: OS is assessed as dead or alive at last follow-up. Tumor response is evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). For target lesions as assessed by MRI or CT: Complete Response (CR) is disappearance of all target and non-target lesions, no new tumors, and normalization of tumor marker level. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions taken as a reference the baseline sum of LDs, and no new tumors. Objective response = CR + PR.
Time Frame: as for outcome 14
Population: Low Risk Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
Participants
  Non-responder and Alive | 79 | 23 | 84
  Non-responder and Dead | 55 | 21 | 84
  Responder and Alive | 21 | 7 | 0
  Responder and Dead | 3 | 3 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC; The null hypothesis that survival is unrelated to objective response versus the alternative hypothesis that objective response is predictive of increased survival for low risk participants receiving LI + CIZ + SOC; Test type: Superiority; p = 0.0101, Fisher Exact
Statistical Analysis 2: Comparison: LI + SOC; The null hypothesis that survival is unrelated to objective response versus the alternative hypothesis that objective response is predictive of increased survival for low risk participants receiving LI + SOC; Test type: Superiority; p = 0.4843, Fisher Exact
Statistical Analysis 3: Comparison: LI + CIZ + SOC vs LI + SOC; Test type: Superiority; p < 0.0067, Fisher Exact — The null hypothesis is that survival is unrelated to objective response versus the alternative hypothesis that objective response is predictive of increased survival for participants receiving LI, considering both treatment groups combined

16. Post Hoc Outcome: Overall Survival by Objective Response (CR+PR) in Low Risk Subjects
Description: OS is assessed using Kaplan-Meier life-table using an unstratified log rank test and a stratified log rank test, stratified by tumor stage, tumor location, and geographic region. Alive at last follow-up was was censored.
  Tumor response is evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). For target lesions as assessed by MRI or CT: Complete Response (CR) is disappearance of all target and non-target lesions, no new tumors, and normalization of tumor marker level. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions taken as a reference the baseline sum of LDs, and no new tumors. Objective response = CR + PR.
Time Frame: as for outcome 14
Population: Low risk Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
Number analyzed (Participants) | 158 | 54 | 168
participants
  Non-responder and Alive | 79 | 23 | 84
  Non-responder and Dead | 55 | 21 | 84
  Responder and Alive | 21 | 7 | 0
  Responder and Dead | 3 | 3 | 0
Statistical Analysis 1: Comparison: LI + CIZ + SOC vs LI + SOC; Null hypothesis is that the Hazard Ratio (HR) for low risk subjects responding to LI (combined arms LI + CIZ + SOC, LI + SOC) is >=1.0 versus the alternative hypothesis that subjects responding to LI are at reduced risk of death (HR < 1.0); Test type: Superiority; p = 0.0131, Regression, Cox; Hazard Ratio (HR) = 0.348, 95% CI 2-sided [0.152 to 0.801]
Statistical Analysis 2: Comparison: LI + CIZ + SOC; Null hypothesis is that the Hazard Ratio (HR) for low risk subjects responding to LI + CIZ + SOC is >=1.0 versus the alternative hypothesis that subjects responding to LI + CIZ + SOC are at reduced risk of death (HR < 1.0); Test type: Superiority; p = 0.0181, Regression, Cox; Hazard Ratio (HR) = 0.246, 95% CI 2-sided [0.077 to 0.787]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of informed consent to the end of the study treatment follow-up. Participants were followed through 60 days after the last radio/chemoradiotherapy. Median last day of radiation-only was 122 days (IQR 106, 132 days). Median last day of chemotherapy for participants receiving both radiation and chemotherapy was 112 days (IQR 96, 129 days). Median AE follow-up was approximately six months post radiotherapy/chemoradiotherapy.
Description: All-cause mortality reports 462 deaths in the ITT population (at risk N=923). All-cause mortality includes the 5 deaths for the 44 subjects excluded from the safety population because they were not treated in this study.
  Adverse events were reported for the safety population (at risk N=879). Five (5) deaths are reported in all-cause mortality that are not reported in the adverse event module.
Arm/Group | LI + CIZ + SOC | LI + SOC | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 204/395 | 68/134 | 190/394
Serious Adverse Events (participants affected / at risk) | 216/383 | 70/129 | 187/367
Other Adverse Events (participants affected / at risk) | 354/383 | 124/129 | 352/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LI + CIZ + SOC (N=383) | LI + SOC (N=129) | Standard of Care (SOC) (N=367)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 100 | 32 | 74
Lip and/or oral cavity cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 6 | 18
Death (General disorders) | 18 | 4 | 17
Pneumonia (Infections and infestations) | 9 | 2 | 11
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 9
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2 | 5
Oral cavity fistula (Gastrointestinal disorders) | 6 | 1 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 2 | 4
Cellulitis (Infections and infestations) | 5 | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 5
Sepsis (Infections and infestations) | 4 | 1 | 3
Cardiac arrest (Cardiac disorders) | 2 | 2 | 3
Postoperative wound infection (Infections and infestations) | 2 | 1 | 4
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1 | 2
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4
General physical health deterioration (General disorders) | 0 | 0 | 5
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 3 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 2
Sudden death (General disorders) | 0 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Tongue cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Abscess neck (Infections and infestations) | 2 | 0 | 1
Wound infection (Infections and infestations) | 2 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Completed suicide (Psychiatric disorders) | 3 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 2 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 2 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 1
Tongue movement disturbance (Gastrointestinal disorders) | 1 | 1 | 0
Tongue necrosis (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Complication associated with device (General disorders) | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 2 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal compression (Gastrointestinal disorders) | 1 | 0 | 0
Oral mucosal hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0
Oroantral fistula (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Submaxillary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Accidental death (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Implant site ulcer (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Organ failure (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ludwig angina (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Flap necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin flap necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin graft contracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epiglottic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lip and/or oral cavity cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Lymphorrhoea (Vascular disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LI + CIZ + SOC (N=383) | LI + SOC (N=129) | Standard of Care (SOC) (N=367)
Anaemia (Blood and lymphatic system disorders) | 64 | 26 | 68
Leukopenia (Blood and lymphatic system disorders) | 36 | 12 | 32
Neutropenia (Blood and lymphatic system disorders) | 33 | 8 | 36
Constipation (Gastrointestinal disorders) | 29 | 9 | 22
Dry mouth (Gastrointestinal disorders) | 40 | 11 | 48
Dysphagia (Gastrointestinal disorders) | 48 | 17 | 40
Nausea (Gastrointestinal disorders) | 38 | 16 | 34
Oral pain (Gastrointestinal disorders) | 31 | 18 | 32
Stomatitis (Gastrointestinal disorders) | 50 | 22 | 63
Vomiting (Gastrointestinal disorders) | 29 | 14 | 24
Asthenia (General disorders) | 29 | 16 | 39
Mucosal inflammation (General disorders) | 121 | 43 | 117
Pyrexia (General disorders) | 43 | 16 | 36
Incision site pain (Injury, poisoning and procedural complications) | 31 | 13 | 37
Radiation injury (Injury, poisoning and procedural complications) | 47 | 13 | 49
Radiation mucositis (Injury, poisoning and procedural complications) | 28 | 15 | 30
Radiation skin injury (Injury, poisoning and procedural complications) | 71 | 31 | 77
Blood creatinine increased (Investigations) | 27 | 8 | 25
Lymphocyte count decreased (Investigations) | 23 | 6 | 26
Weight decreased (Investigations) | 169 | 56 | 168
Decreased appetite (Metabolism and nutrition disorders) | 18 | 7 | 21
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 | 13 | 11
Insomnia (Psychiatric disorders) | 25 | 5 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 4 | 17
Dermatitis (Skin and subcutaneous tissue disorders) | 48 | 12 | 43
Scar pain (Skin and subcutaneous tissue disorders) | 28 | 7 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
See Clinical Protocol Section 13.0 Publication Plan

DOCUMENTS (7):
  • Study Protocol (2014-06-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/Prot_000.pdf
  • Statistical Analysis Plan: SAP main text (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_001.pdf
  • Statistical Analysis Plan: CS001P3 Note to File 1 (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_002.pdf
  • Statistical Analysis Plan: CS001P3 Note to file 2 (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_003.pdf
  • Statistical Analysis Plan: Note to file 3 (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_004.pdf
  • Statistical Analysis Plan: Note to file 4 (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_005.pdf
  • Statistical Analysis Plan: Note to file 5 (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT01265849/SAP_006.pdf